CLINICAL TRIAL: NCT01721590
Title: Study of Tongxinluo to Improve High on Clopidogrel Platelet Reactivity in Patients With Coronary Heart Disease
Brief Title: Tongxinluo Improve High on Clopidogrel Platelet Reactivity Patients With Coronary Heart Disease
Acronym: Talent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Han Yaling (Other)
Responsible Party: Sponsor-Investigator, Han Yaling, vice president, Shenyang Northern Hospital
Organization: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYNH-20120929
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: high on-treatment platelet reactivity; Coronary Heart Disease; Tongxinluo
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — tongxinluo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Placebo，3 capsules/time，3times/day for 1 year
  Interventions: Drug: placebo
- Tongxinluo (Experimental): Tongxinluo 3 capsules/time 3times/day for 1 year
  Interventions: Drug: Tongxinluo

INTERVENTIONS:
Drug: Tongxinluo — Tongxinluo,3 capsules/time 3times/day for 1 year
  Other Names: Tongxinluo capsule
  Arms: Tongxinluo
Drug: placebo — 3 capsules/time，3times/day for 1 year
  Other Names: placebo capsules
  Arms: Control

SUMMARY:
Tongxinluo is a kind of Chinese patent drug,which could promote blood circulation.Recent reports suggested that tongxinluo's effectiveness in reducing the thrombin activity.In this prospective randomized study,all patients in control group will receive blank placebo ,all patients in test group will receive tongxinluo.All patients will be followed up for one year.

DETAILED DESCRIPTION:
The primary endpoint is Platelet Reaction Unit( by VerifyNow) at 30 days.The secondary endpoints include inflammation marker (hsCRP、CD62P-CD41),TT,FIB and PT at 30 days,and MI、Ischemic Stroke, target vessel revascularization and all-cause mortality 、bleeding events at 1 year.

ELIGIBILITY:
Inclusion Criteria:

- (1)ACS (including unstable angina pectoris, non-ST-segment elevation myocardial infarction and ST-elevation myocardial infarction) （2）Accept at least one coronary stent. （3）The age between18 and 75 . （4）High on-treatment platelet reactivity defined as an ADP-induced platelet aggregation (by VerifyNow，PRU≥236）at 24 hr after clopidogrel loading (300 ~ 600mg)or 24 hours after PCI.

（5）Informed Consent

Exclusion Criteria:

* （1）Tongxinluo contraindication . （2）Receiving GP IIb / IIIa receptor antagonist treatment （3）Who complicate the known bleeding tendency and blood system diseases. （4）NYHA grade III ~ IV （5）Aspirin or clopidogrel allergies （6）Severe liver or kidney dysfunction （7）Pregnancy （8）Cann't accept 30 days supervision and blood proofer. （9）Other serious illness, life expectancy less than 6 months. （10) Planned surgery recently （11) PCI again within 30 days. (12) Mental diseases interfering understanding the informed consent form （13）Accept other drugs or participate in other clinical research at the same time .

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Platelet reaction unit(PRU) measured by verifyNow | 1 month
  to measure the rate of HPR(PRU ≤ 235)

SECONDARY OUTCOMES:
Inflammation Marker (hsCRP、CD62P-CD41) | 1 month
Plasma fibrinogen concentration | 1 month
Thrombin time | 1 month
Prothrombin time | 1 month
major adverse cardiovascular events | 1 year
  Including MI,Stroke,target vessel revascularization,and all-cause mortality
bleeding event | 1 year
Adverse drug reaction and withdrawal rate | 1 month ，1 year
Angina recurrence | 1 year
Traditional Chinese medicine angina symptoms scores | 1 year
Intra-stent thrombosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Dr, Principal Investigator — Shenyang Northern Hospital
Locations (3):
- China (3):
  - ShenZhou Hopital Of ShenYang Medical College, ShengYang, Liaoning
  - The 463th Hospital Of PLA, Shenyang, Liaoning
  - Northern Hospital, Shenyang, Liaoning